CLINICAL TRIAL: NCT01121757
Title: A Phase 2 Study Evaluating the Efficacy of Epigenetic Modulation in Relapsed/Refractory Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: Epigenetic Modulation in Relapsed/Refractory Follicular Lymphoma and Marginal Zone Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed temporarily in February 2012 pending analysis of samples collected. In October, 2012, Celgene requested closure of the study.
Sponsor: Duke University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019069
Record Dates: First submitted 2010-02-11; First posted 2010-05-12 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: relapsed; refractory; lymphoma; follicular; marginal zone
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Recurrence; Lymphoma | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azacitidine followed by Lenalidomide (Experimental): Azacitidine 75 mg/m2 subcutaneously (SC) or IV on days 1-5; subjects will begin Part 2 at the azacitidine dose level tolerated in Part 1a.
  Lenalidomide dose is 15mg po per day on days 1-21; starting dose during Part 2 will depend upon how well the subject tolerated drug during Part 1.
  Interventions: Drug: azacitidine; Drug: lenalidomide
- Lenalidomide followed by Azacitidine (Experimental): Lenalidomide dose is 15mg po per day on days 1-21; starting dose during Part 2 will depend upon how well the subject tolerated drug during Part 1.
  Azacitidine 75 mg/m2 subcutaneously (SC) or IV on days 1-5; subjects will begin Part 2 at the azacitidine dose level tolerated in Part 1a.
  Interventions: Drug: azacitidine; Drug: lenalidomide

INTERVENTIONS:
Drug: azacitidine — Azacitidine 75 mg/m2 SC or IV on days 1-5; subjects will begin Part 2 at the azacitidine dose level tolerated in Part 1a.
  Other Names: Vidaza
Drug: lenalidomide — Lenalidomide dose is 15mg po per day on days 1-21; starting dose during Part 2 will depend upon how well the subject tolerated drug during Part 1.
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to evaluate the response and safety in subjects receiving the drugs lenalidomide and azacitidine when each drug is given by itself and when the drugs are taken together. This study is open for patients with relapsed or refractory follicular or marginal zone lymphoma.

DETAILED DESCRIPTION:
This will be a prospective, non-randomized, un-blinded, phase 2 efficacy trial using an Immunomodulatory derivatives of thalidomide (IMiD™)compound and a hypomethylating agent for epigenetic targeted therapies in patients with relapsed/refractory follicular and marginal zone lymphoma. There will be two parts to the trial. Each patient will progress through each part of the study.

Part 1: Sequential single agent therapy with azacitidine and lenalidomide. Each agent will be given for four-six 28-day cycles.

Subjects with less than a complete response (CR) after 4 cycles of study drug in Part 1a or 1b should proceed to the next study drug(s) after the prescribed washout period.

Subjects with a CR may receive up to 6 cycles of study drug and will not receive the next study drug(s) until there is evidence of progressive disease.

There will be a 1-6 week 'washout' period between stopping and starting each agent in Part 1, unless rapid progression suggests holding therapy would not be in the patient's best interest. There will be no washout period required between Part 1 and Part 2.

Part 2: Combination therapy with azacitidine and lenalidomide given in 28-day cycle for up to 13 cycles in subjects who have stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Follicular or Marginal Zone Lymphoma
2. Refractory disease defined as persistence of evaluable disease after therapy or have relapsed disease to at least one prior treatment regimen
3. Understand and voluntarily sign an informed consent form
4. Age > or = to 18 years
5. Able to adhere to the study requirements
6. A frozen tumor sample must be available for microarray analysis. This may either be a previously collected sample if it was properly prepared or a new biopsy may be obtained.

   o At least 1 core biopsy specimen using at least a 16 gauge needle, which corresponds to roughly 25 mg of tissue. An equivalent amount of biopsy material from previously performed procedures, as long as it was fresh frozen, can be used. Sample obtained with leukapheresis is acceptable in subjects with a white blood cell count (WBC) of 100,000 or greater.
7. Eastern Cooperative Oncology Group (ECOG) performance status of < or = to 2
8. Laboratory test results within ranges specified by the protocol.
9. Disease free of prior malignancies for > or = to 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast or superficial melanoma only requiring excision or prostate cancer with a prostate specific antigen (PSA) that has not increased for at least 3 months.
10. All study participants must be willing to be registered into the mandatory RevAssist® program, and comply with the requirements of RevAssist®.
11. Females of childbearing potential (FCBP) must comply with pregnancy testing requirements. Men and women must use approved birth control methods during the study.
12. Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with azacitidine.
13. If at high risk for thrombotic event (such as on steroids or history of deep vein thrombosis), subjects must be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid may use warfarin or low molecular weight heparin)

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide or mannitol.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
7. Any prior use of lenalidomide or azacitidine
8. Concurrent use of other anti-cancer agents or treatments
9. Known positive for HIV or infectious hepatitis, type B or C
10. No chemotherapy, biologics or immunotherapy within 2 weeks prior to registration as specified in the protocol. Subjects must have recovered from all therapy-related non-hematological toxicities to < grade 1 or to baseline if patient started with > grade 1 toxicity. There is no time limit with regards to radiation prior to registration.
11. No radioimmunotherapy within 2 months prior to registration. Subjects must have recovered from all therapy-related toxicities to < grade 1 or to baseline if patient started with > grade 1 toxicity.
12. No prior allogeneic stem cell transplantation unless allogeneic engraftment is <2%
13. Subjects receiving chronic, systemic treatment with corticosteroids equivalent to >20mg of prednisone per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne W. Beaven, MD, Principal Investigator — Duke University Medical Center Durham, NC USA
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 2010 through January 2012 from the Duke Cancer Institute.
Pre-assignment Details: The first 3 patients started on 1a and the next 3 patients started in 1b and the next 3 were in 1a and so on. Eleven subjects consented to the study, 1 patient elected other treatment options prior to assignment and 1 other patient converted to Diffuse Large B-Cell Lymphoma, which made them ineligible.
Groups:
- 1a-Azacitidine Followed by Lenalidomide: Subjects will take azacitidine for 4-6 cycles (first drug) followed by a 1-6 week washout period. Subjects with a Complete Remission (CR) may receive up to 6 cycles of first drug and will not receive the next until disease progression.
  Subjects with less than a CR after 4 cycles of azacitidine (first drug) will proceed to receive lenalidomide (second drug) for 4-6 cycles.
  Subjects with a CR after lenalidomide may receive up to 6 cycles of lenalidomide and will not start on the combination drug until disease progression.
  The combination therapy (azacitidine and lenalidomide) will be given in 28-day cycles for up to 13 cycles in subjects who have stable disease or better.
- 1b-Lenalidomide Followed by Azacitidine: Subjects will take lenalidomide for 4-6 cycles (first drug) followed by a 1-6 week washout period. Subjects with a Complete Remission (CR) may receive up to 6 cycles of first drug and will not receive the next until disease progression.
  Subjects with less than a CR after 4 cycles of lenalidomide (first drug) will proceed to receive azacitidine (second drug) for 4-6 cycles.
  Subjects with a CR after azacitidine may receive up to 6 cycles of azacitidine and will not start on the combination drug until disease progression.
  The combination therapy (azacitidine and lenalidomide) will be given in 28-day cycles for up to 13 cycles in subjects who have stable disease or better.
Period: First Drug
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Started | 6 | 3
Completed | 5 (Completed a minimum of 4 cycles of Azacitidine.) | 1 (Completed a minimum of 4 cycles of Lenalidomide)
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Disease Progression | 0 | 2
Period: Second Drug
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Started | 4 (1 subject did not start drug 2 due to disease progression) | 1
Completed | 4 | 1
Not Completed | 0 | 0
Period: Combination
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Started | 2 (2 subjects did not start combination drug. 1 elected surgery 1 had a complete response after drug 2.) | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Disease Progression | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Predicted by Molecular Signatures Compared to True Response
Description: The predicted response (response to therapy vs. no response to therapy) using gene sequencing will be compared to the overall "true" response (reported in Primary Outcome 2).
Time Frame: approximately one year
Population: The number of participants who were evaluated for a response were analyzed to see if the prediction of response vs. no response through gene expression matched the true response.
Measure: Number; unit: participants
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Number analyzed (Participants) | 6 | 3
participants
  Predicted: Response; Actual: Response | 1 | 0
  Predicted: No Response; Actual: No Response | 2 | 3
  Predicted: Response; Actual: No Response | 3 | 0

2. Primary Outcome: Overall Response
Description: Number of patients with a complete or partial response using Cheson criteria for lymphoma.
  A complete response is defined as a complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy. A partial response is defined as a greater than or equal to 50% decrease in the sum of the products of the greatest diameters of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Patients who have been on study drug for at least 2 months will be considered evaluable for response as long as they have had repeat imaging to assess response or clear progression based on physical exam.
Time Frame: Response will be assessed after at least 4 months on first study drug.
Population: Everyone who started the first drug regimen
Measure: Number; unit: participants
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Number analyzed (Participants) | 6 | 3
participants | 1 | 0

3. Primary Outcome: Overall Response
Description: as for outcome 2
Time Frame: Response will be assessed after at least 4 months on second drug.
Population: Everyone who started the second drug regimen
Measure: Number; unit: participants
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Number analyzed (Participants) | 4 | 1
participants | 2 | 0

4. Primary Outcome: Overall Response
Description: as for outcome 2
Time Frame: Response will be assessed after at least 6 months on combination drug.
Population: Only subjects that completed combination drug will be included in analysis.
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Grade 3 and 4 Toxicities
Description: Evaluate the safety of lenalidomide, azacitidine and the combination of azacitidine + lenalidomide in patients with lymphoma; grading the adverse events using Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: While taking the study drug and 30 days after the last dose
Measure: Number; unit: participants
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Number analyzed (Participants) | 6 | 3
participants
  Grade 3 | 5 | 3
  Grade 4 | 1 | 1

6. Other Pre Specified Outcome: Serum Markers Measured on the First Day of Cycle 1 and on the First Day of Cycle 3
Time Frame: Within 4 months of taking single agent and 6 months of taking the combination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: We collect adverse event information from the time they start drug until 30 days after the last dose.
Arm/Group | 1a-Azacitidine Followed by Lenalidomide | 1b-Lenalidomide Followed by Azacitidine
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1a-Azacitidine Followed by Lenalidomide (N=6) | 1b-Lenalidomide Followed by Azacitidine (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis (left lower extremity) (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Breast Cancer) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Cecal adenocarcinoma ) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Refractory Anemia with Excess blasts-1) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1a-Azacitidine Followed by Lenalidomide (N=6) | 1b-Lenalidomide Followed by Azacitidine (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (8) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colonic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (13) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Spasms) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (7) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 6 (8) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Herpes Zoster) (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Right 5th finger) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (5) | 0 (0)
Neutropenia (Investigations) | 4 (6) | 0 (0)
Thrombocytopenia (Investigations) | 2 (10) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (4) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (4) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Paresthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (8) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (10) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes